CLINICAL TRIAL: NCT07227649
Title: NAC-REPAIR: N-Acetylcysteine-facilitated Redox-Immune Modulation for Post-surgical Analgesia and Injury Recovery
Brief Title: NAC-REPAIR for Post-surgical Pain
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Banner University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00007009
Record Dates: First submitted 2025-11-10; First posted 2025-11-13 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Carpal Tunnel Surgery; Trigger Finger Disorder; De Quervain Syndrome; Guyon's Canal; Dupuytren Contracture; Morton Neuroma; Tarsal Tunnel Syndrome; Plantar Fasciopathy; Peroneal Nerve Entrapment
MeSH Terms: conditions — Trigger Finger Disorder; Dupuytren Contracture; Morton Neuroma; Tarsal Tunnel Syndrome; Peroneal Neuropathies

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- N-Acetylcysteine (NAC) (Experimental): Intervention: Oral N-acetylcysteine capsules, 600 mg twice daily.
  Timing/Duration: Begin the evening before surgery (≤24 h pre-op) and continue through Post-op Day 14 (total 15 days; bottle overfilled to cover missed doses).
  Administration: Self-administered at home; counseling at baseline dispense; pill diary + pill counts.
  Concomitant care: All peri-operative care per standard of care (SoC), including multimodal analgesia; no high-dose antioxidant supplements; nitrates excluded.
  Objective: Test whether peri-operative NAC improves early pain, function, and recovery via redox-immune modulation.
  Interventions: Drug: NAC
- Placebo (Placebo Comparator): Intervention: Matched inert capsules (e.g., microcrystalline cellulose), identical in size/appearance/labeling to NAC.
  Timing/Duration: 600 mg-equivalent capsule count, twice daily, evening before surgery through Post-op Day 14.
  Administration: Same counseling, diary, and adherence checks as NAC arm.
  Concomitant care: Identical SoC allowances/restrictions as NAC arm.
  Interventions: Drug: NAC 0mg/day (Placebo)

INTERVENTIONS:
Drug: NAC — Intervention: Oral N-acetylcysteine capsules, 600 mg twice daily.
  Timing/Duration: Begin the evening before surgery (≤24 h pre-op) and continue through Post-op Day 14 (total 15 days; bottle overfilled to cover missed doses).
  Administration: Self-administered at home; counseling at baseline dispense; pill diary + pill counts.
  Concomitant care: All peri-operative care per standard of care (SoC), including multimodal analgesia; no high-dose antioxidant supplements; nitrates excluded.
  Objective: Test whether peri-operative NAC improves early pain, function, and recovery via redox-immune modulation.
  Arms: N-Acetylcysteine (NAC)
Drug: NAC 0mg/day (Placebo) — Intervention: Matched inert capsules (e.g., microcrystalline cellulose), identical in size/appearance/labeling to NAC.
  Timing/Duration: 600 mg-equivalent capsule count, twice daily, evening before surgery through Post-op Day 14.
  Administration: Same counseling, diary, and adherence checks as NAC arm.
  Concomitant care: Identical SoC allowances/restrictions as NAC arm.
  Randomization/Blinding: 1:1, stratified by surgery type (upper- vs lower-extremity); double-blind (participants, investigators, assessors).
  Primary comparisons: Early postoperative pain and function (e.g., PROMIS-PI/PF, QuickDASH or LEFS), opioid consumption; safety/tolerability.
  Arms: Placebo

SUMMARY:
This pilot asks whether peri-operative N-acetylcysteine (NAC) improves recovery after common outpatient hand/foot-ankle surgery-specifically, does NAC reduce pain and opioid use and enhance function by modulating redox-inflammatory pathways? Primary objectives are to establish feasibility (accrual, adherence, follow-up), estimate NAC vs placebo effects on pain, function, and opioid consumption, and characterize inflammatory signatures that may predict response.

Methods: a single-site, double-blind, 1:1 randomized trial (N≈80) comparing NAC 1,200 mg twice daily for 14 days (starting pre-op) vs matching placebo; daily e-diaries for POD0-14; standardized outcomes (PROMIS Pain Interference; QuickDASH or FAAM; PGIC; opioid MME); and small blood draws pre-surgery and at two follow-up visits for cytokine profiling.

ELIGIBILITY:
Inclusion Criteria:

* Elective outpatient hand/upper-extremity or foot/ankle surgery (single site; same-day discharge)
* Baseline visit feasible ≤14 days pre-op
* Can complete surveys/blood draw
* Provides informed consent
* Willing to follow dosing schedule and avoid restricted supplements/meds

Exclusion Criteria:

* Allergy to NAC/capsule components □ NAC or high-dose antioxidants in past 14 days (unwilling to stop)
* Chronic daily opioids ≥3 months or OUD/maintenance therapy □ Pregnant/breastfeeding or no contraception as applicable
* Daily nitrates (nitroglycerin/isosorbide) □ Planned >24h admission, multistage/trauma case □ Other interventional study within 30 days
* Unable to swallow capsules / malabsorption surgery affecting oral meds

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
PROMIS pain interference | baseline; post-op (2-4 weeks); post-op (12 weeks);
  Patient-Reported Outcomes Measurement Information System - Pain Interference T-score metric: mean = 50, SD = 10 Higher scores = worse outcome (greater pain interference with daily activities, social, cognitive, emotional, and physical functioning)

SECONDARY OUTCOMES:
PROMIS Physical Function | Baseline; post-op (2-4 weeks); post-op (12 weeks)
  Patient-Reported Outcomes Measurement Information System Physical Function T-score metric: mean = 50, SD = 10 Higher scores = better outcome (greater ability to carry out physical activities such as mobility, self-care, and instrumental activities)
Numeric Pain Rating Scale | Baseline; post-op (2-4 weeks); post-op (12 weeks)
  0-10: 0 = no pain, 10 = worst imaginable Higher scores = worse outcome (greater perceived pain intensity)

CONTACTS AND LOCATIONS:
Locations (1):
- Banner Health, Tucson, Arizona, United States